CLINICAL TRIAL: NCT01601249
Title: A Prospective Comparison Between Conventional IVF Embryo Grading and Polscope Based Grading
Brief Title: Improving IVF Embryo Quality Grading Using Polarized Light
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: PI moved from Hadassah
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 008212- HMO-CTIL
Record Dates: First submitted 2012-05-03; First posted 2012-05-17 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2012-05

CONDITIONS: Infertility
Keywords: IVF, embryo selection, polarized light
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Polscope based embryo grading (Experimental): Embryos for transfer will be selected based on highest polscope scores, unless are not grade 1-2 by conventional morphology
  Interventions: Procedure: Embryo selection based on polscope grading or morphology
- Morphology based embryo grading (Active Comparator): Conventional embryo grading and decision making
  Interventions: Procedure: Embryo selection based on polscope grading or morphology

INTERVENTIONS:
Procedure: Embryo selection based on polscope grading or morphology — In the experimental arm embryo grading will be performed by polscope rather than conventional morphology, and the best embryo/s for transfer will be selected by this method.

SUMMARY:
Selecting one or two IVF embryos with the highest potential to implant is extremely important for the success of the treatment- obtaining pregnancies and avoiding multi-fetal gestations. The currently used IVF embryo grading method is based solely on embryo morphology (cleavage rate and fragmentation) just before the transfer, which is not very well correlated with the implantation potential of each embryo. Oocyte quality and adequacy are the most important factors determining the biological quality and implantation potential of the embryo. It impossible to grade oocytes using plain optical systems, other than maturity and gross anomalies.

Polscope systems allow to visualize intra ooplasmic structures and determine their retardance, as well as that of the Zona Pellucida. The investigators hypothesize that grading embryos using the oocyte's parameters as visualized by polscope is superior to conventional morphology and correlates better with their implantation potential.

Here the investigators will perform a prospective randomized controlled trial to examine this hypothesis.

DETAILED DESCRIPTION:
Each embryo will be graded in accordance to polscope based parameters; the presence of a spindle in the oocyte, its retardance, the distance between the spindle and the PB, and the thickness and retardance of the ZP.

In the experimental group the embryos for transfer will be selected based on these parameters, whereas in the control group they will be selected based on conventional morphologic criteria.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-38, (near) normal MF, normal uterus, >4 aspirated oocytes, intent to transfer 1-2 embryos.

Exclusion Criteria:

* Severe MF problems, uterine anomalies, PGD, RIF.

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2012-09; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Occurrence of clinical pregnancy | within 2 weeks after ET

SECONDARY OUTCOMES:
Live birth | up to 40 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yoel Shufaro, MD PhD, Principal Investigator — HMO
Locations (1):
- Hadassah University Hospital, Jerusalem, Israel